CLINICAL TRIAL: NCT04407793
Title: Prospective and Multicentre Study on Clinical-biological Factors Predictive of Chronic Colon DIverticulitis
Acronym: DICRO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sebastiano Biondo (Other)
Responsible Party: Sponsor-Investigator, Sebastiano Biondo, Sebastiano Biondo. Clinical Professor. Head of Surgery Department, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Other Study IDs: DICRO-2020
Record Dates: First submitted 2020-05-25; First posted 2020-05-29 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Acute Diverticulitis
Keywords: Acute diverticulitis; Chronic diverticulitis; Recurrence; Diverticulitis treatment
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Faecal samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Diverticulitis Group: Patients with acute diverticulitis episode
- Diverticulosis group: Patients diagnosed with diverticulosis without any acute diverticulitis episode
- Non-diverticulosis: Patients without diverticulosis

SUMMARY:
MAIN OBJECTIVE: Description of predicted markers of acute diverticulitis crisis, using bivariate and multivariate analyses. Analysis of acute diverticulitis predictor swings.

SIDE OBJECTIVES: Descriptive analysis of HRQL in the different measurement periods to establish the evolution of the disease. Correlate HRQL values of systemic and local inflammatory markers in the diverticulitis group. Sub-analysis of patients with immunosuppression to evaluate disease virulence compared to a group of patients without immunosuppression.

STUDY TYPE: Clinical, observational, prospective and multicenter study (8 hospitals) with three study groups: patients diagnosed with acute diverticulitis attending emergencies, diverticulosis patients and patients without diverticulums. INCLUSION CRITERIA: Age > 18years and radiological diagnosis by abdominal CT acute diverticulitis. EXCLUSION CRITERIA: Rejection of the patient -severe diverticulitis requiring urgent surgery -an inability to understand HRQL questionnaire - IBD - pregnancy or breastfeeding - acute diverticulitis within the prior year of the study - Roma IV criteria fulfilment. VARIABLES: Main variables: local and systemic inflammatory markers- faecal calprotectin. Secondary variables: recurrence of acute diverticulitis -the persistence of symptoms - SF 12 and GIQLI questionnaires.

STATISTICS: Sample size: alpha error 0.05; beta error 0.20; bilateral; proportion 0.9 in the control group; 500 subjects group diverticulitis, 200 group diverticulosis and not diverticulums.

DETAILED DESCRIPTION:
GENERAL CHARACTERISTICS OF THE PROJECT:

Despite being a benign pathology, colon diverticulitis represents the fifth most important gastrointestinal pathology and has a great clinical impact on the quality of life of patients and on health expenditure. Understanding a disease involves being able to make the correct diagnosis of the patient and most importantly for the patient, an adequate treatment of his symptoms. It is required to give accurate information to the patient and answer his doubts, although the pathophysiology of the disease is unknown. As it is a benign disease with heterogeneous behaviours and manifestations, it is difficult to make the decision related to undergo surgery. This decision could be facilitated if it is based on extensive information from the doctor. It is also important to be able to select those patients who have a higher risk of relapse in order to prioritize them on the waiting list for surgery. As a benign disease with occupational active patient involvement, acute diverticulitis has a major economic impact by leading to repeat leaves in some patients, who are even on a waiting list to operate.

EXPECTED IMPACT:

We believe that this project can respond to the management of a group of patients, in which there is currently no consensus in the Scientific Community. Therefore, our results are transferable, as we intend to establish the pathophysiology of the entity known as chronic diverticulitis and detect the predictors of that entity. Currently, there is no consensus on the therapeutic management of patients with recurrent episodes of diverticulitis or persistent symptoms, so that they are treated differently at the discretion of the surgeon, without any scientific basis. It is also unclear whether it is a maintained inflammatory disorder or a functional disorder, which differentiation is basic in order to indicate a correct treatment of the patients. In addition, there is an information gap, unable to respond if a patient with acute diverticulitis will have a high or low probability of recurrence and at what time. There are still no studies answering these questions, key to choosing the best treatment and to give an answer to the huge population of diverticulitis patients.

HYPOTHESIS.

1. Establish a therapeutic algorithm in patients diagnosed with acute diverticulitis who go to the emergency department, whose initial management is not an urgent surgical intervention.
2. There is an inflammatory physiopathology underlying between acute episodes, which can play a role in the apparition of the new episode of acute diverticulitis.

OBJECTIVES:

* Description of prognostic factors of new episodes of acute diverticulitis which can be easy detected in the outpatient clinic, and creation of a therapeutic algorithm that allows selecting patients who could benefit from early surgery
* Descriptive analysis of symptoms with Health Related Quality of Life questionnaires (HRQL), in order to establish the evolution of the disease and correlate symptoms with systemic and local inflammatory markers.
* Sub-analysis of patients with immunosuppression to assess the virulence of the disease.

METHODOLOGY RECRUITMENT. All patients who meet the inclusion criteria, do not present any exclusion criteria and voluntarily agree to participate in the study after having been visited and diagnosed in the following hospitals will be included: Bellvitge University Hospital (Barcelona), Vall d 'University Hospital Hebron (Barcelona), University Hospital del Mar (Barcelona), Moises Broggi University Hospital (Barcelona), Joan XXIII University Hospital (Tarragona), Parc Taulí University Hospital (Sabadell), Althaia Hospital (Manresa), Josep Trueta University Hospital (Girona). All patients will receive an information sheet and informed consent. Once the patients are considered eligible and have formulated their questions and/or doubts to the investigator, they will be included.

STUDY GROUP (1): Patients with acute diverticulitis who come to the emergency department. It will be taken in the emergency department Blood tests that include leukocyte count and formula, C-reactive protein, Neutrophil-Lymphocyte ratio calculation, Platelet-lymphocyte ratio, lymphocyte-monocyte ratio, Modified Glasgow Prognostic Score. Faecal calprotectin (the collection tube that the patient must deliver after the first deposition will be delivered).

FOLLOW-UP:

1. all patients included in the study as DIVERTICULITIS GROUP, at the month of episode 3, 6, 12, 18 and 24 months of the first episode with Blood analysis with detection of inflammatory systemic markers that will include leukocyte count, leukocyte formula, Protein- C reactive. Neutrophil-Lymphocyte ratio, Platelet-lymphocyte ratio, lymphocyte-monocyte ratio, Modified Glasgow Prognostic Score. Faecal calprotectin Delivery to the patient of the stool sample collection kit. It will be delivered within 7 days, HRQL Questionnaires (SF-36) at 3, 6, 12, 18 and 24 months after the first episode of acute diverticulitis. They will be delivered in the outpatient clinic. Colonoscopy at 2 months after the first episode. It will be requested on the first month's post-diverticulitis visit when the informed consent will be signed. In the colonoscopy, the following will be analyzed: endoscopic description based on a description of the endoscopic mucosa. Sampling and sending to the organizing centre of the project (Bellvitge University Hospital): Sample A: 1-5cm of diverticulum that has participated in diverticulitis episode Sample B: 30cm of the area that has suffered diverticulitis. Rome VI criteria at 3 months follow-up. Sampling for the study of local inflammatory markers: IL-6, IL-10, tumour necrosis factor (TNF), macrophages, calculation of inflammation index of Ulcerative Colitis. All data will be collected in the workbook-CRD website.
2. DIVERTICULOSIS GROUP AND CONTROL GROUP: Patients with asymptomatic diverticula and patients without diverticula. DIVERTICULOSIS GROUP. Samples will be collected from patients undergoing colonoscopy for another reason (polyp control) and diagnosed with diverticulosis, without having presented an episode of recent diverticulitis.

Only patients from the organizing centre (Bellvitge University Hospital) will be included.

CONTROL GROUP. Patients who undergo colonoscopy for another reason (polyps control) and no diverticulosis is found. Only patients from the organizing centre (Bellvitge University Hospital) will be included. Test to take: A blood test that will include leukocyte count and leukocyte formula, C-reactive protein. Neutrophil-Lymphocyte ratio], Platelet-lymphocyte ratio, lymphocyte-monocyte ratio, Modified Glasgow Prognostic Score. Faecal calprotectin (LOOK ANNEX-protocol for collection and storage of stool sample). Colonoscopy with sample for the study of local inflammatory markers: IL-6, IL10, tumour necrosis factor (TNF), local macrophages: Endoscopic description based on a description of the mucosa Endoscopic Sampling: Sample A: 1-5cm from any diverticulum, if any (diverticulosis group). In case there are no diverticula, 2 random samples, Sample B: 30 cm from the diverticulosis area if any. In case there are no diverticula, 2 random samples. Collection of results in the workbook-CRD website.

DESCRIPTIVE VARIABLES OF THE POPULATION: -Numerical variable of identification of the case -Age-Sex -Previous episodes of acute diverticulitis- Date of the episodes -Consumption of alcohol- Tobacco consumption- exercise.

MAIN VARIABLE. Local and systemic inflammatory markers. Calprotectin.

SECONDARY VARIABLES: Colonoscopy markers -Quality of life questionnaire SF-12/GIQLI - immunosuppression.

SCHEDULE:

* 1)Patient recruitment period: 1 year
* 2)Follow-up of patients: 2 years from the date of the first episode
* 3)Data entry: parallel to the follow-up of patients in the workbooks-CRD website.
* 4)Debugging and data analysis: parallel to the follow-up of patients.
* 5)External monitoring and auditing of the centres one year after the start of data collection, midway through the study and at the end of inclusion.
* 6)Preparation of articles for the publication of the results: 1 year after the process of collection and statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18years
* Current episode of acute diverticulitis diagnosed with abdominal CT

Exclusion Criteria:

* Rejection of the patient
* Severe diverticulitis requiring urgent surgery
* Inability to understand HRQL questionnaires
* IBD background
* Pregnancy or lactation
* Acute diverticulitis episodes within the prior year to the start of the study
* Patients who meet Roma IV criteria for IBS

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: DIVERTICULITIS COHORT: Patients with current acute diverticulitis, diagnosed with abdominal CT and not requiring urgent surgery for this reason
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-05-25 (Actual); Primary Completion 2021-05-25 (Estimated); Study Completion 2023-05-25 (Estimated)

PRIMARY OUTCOMES:
Recurrence of acute diverticulitis | 2 years
  To detect which patients with acute diverticulitis recur
Systemic inflammatory markers | 2 years
  To correlate systemic inflammatory markers with acute diverticulitis recurrence.
  * Systemic inflammatory markers include: A blood test with leukocyte count and formula, C-reactive protein, albumin, Neutrophil-Lymphocyte ratio calculation, Platelet-lymphocyte ratio calculation, lymphocyte-monocyte ratio calculatio, Modified Glasgow Prognostic score calculation.
Faecal calprotectine | 2 years
  To correlate faecal calprotectine with acute diverticulitis recurrence
Local inflammatory markers | 2 years
  To correlate local inflammatory markers with systemic inflammatory markers and recurrence.
  *Local inflammatory markers come from colonic endoscopic samples taken in the colonoscopy at 2 months after the acute diverticulitis episode. 2 samples are taken:
  * Sample A: 1-5cm of diverticulum that has participated in diverticulitis episode (correlated with the CT)
  * Sample B: 30cm of the area that has suffered diverticulitis. Sampling for the study of local inflammatory markers includes IL-6, IL-10, tumour necrosis factor (TNF), macrophages, eosinophils and calculation of inflammation index of Ulcerative Colitis.

SECONDARY OUTCOMES:
HRQL (Health Related Quality of Life) QUESTIONNAIRES | 2 years
  To correlate clinical symptoms with inflammatory markers.
  Questionnaires used:
  * SF-12 Health Survey, in order to measure Mental and Physical Health. There are 8 areas with a minimum value of 0 (the worst health state) and a maximum of 100 (best health state)
  * GIQLI (Gastrointestinal Quality of Life questionnaire). Minimum value of 0 (the worst health state) and a maximum of 100 (best health state)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Bellvitge, Barcelona, Spain

REFERENCES:
- [Derived] Climent M, Sobrino L, Guardiola J, Kreisler E, Biondo S; DICRO Trial Group. Prospective and multicenter study on clinical-biological factors predictive of chronic colon diverticulitis: DICRO Trial. Int J Colorectal Dis. 2025 May 7;40(1):111. doi: 10.1007/s00384-025-04902-0. PMID 40335755